CLINICAL TRIAL: NCT02477709
Title: A Study to Assess the Tolerability of a Single Dose of AF-219, a P2X3 Receptor Antagonist, in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Assess the Tolerability of a Single Dose of Gefapixant (AF-219/MK-7264) in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7264-019; AF219-019 (Other: Afferent Pharmaceuticals)
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Gefapixant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefapixant (Experimental): Gefapixant oral tablets (150 mg) administered as a single dose
  Interventions: Drug: Gefapixant

INTERVENTIONS:
Drug: Gefapixant — Gefapixant oral tablet (150 mg administered as three 50 mg tablets) - single dose only
  Other Names: AF-219; MK-7264

SUMMARY:
This study assesses the tolerability of a single dose of gefapixant (AF-219) in participants with idiopathic pulmonary fibrosis (IPF). Six eligible participants will receive a single 150 mg dose of gefapixant and undergo tolerability and PK assessments.

DETAILED DESCRIPTION:
This study assesses the tolerability of a single dose of gefapixant in participants with idiopathic pulmonary fibrosis (IPF).

This will be the first experience of administering gefapixant in patients with IPF. P2X3 receptors are found on the chemosensory afferents of the carotid body and can influence sympathetic autonomic discharge, especially in sensitized subjects; accordingly, by blocking these P2X3 receptors, gefapixant may have an effect of reducing sympathetic activity. Therefore in order to determine whether P2X3 antagonism would have an effect on the hemodynamic measures such as blood pressure in patients with IPF, study AF219-019 is being performed. These patients will be closely monitored in order to determine any such effect.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic pulmonary fibrosis diagnosis based upon the American Thoracic Society (ATS)/ European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/ Latin American Thoracic Society (ALAT) IPF 2011 guideline
* Life expectancy of greater than 6 months
* Stable medical condition (IPF) for at least 4 weeks
* Women of child-bearing potential must use 2 forms of an acceptable birth control method from Screening through the Follow-Up Visit
* Male subjects and their partners of child-bearing potential must use 2 methods of acceptable birth control, 1 of which must be a barrier method, and make no donation of sperm from Screening until 3 months after the last dose of study drug
* Written informed consent
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Current smoker (i.e., within the last 30 days)
* Initiation of treatment with an antihypertensive agent within 4 weeks prior to the day of dosing (Day 1) or during the study
* History of upper respiratory tract infection within 4 weeks of the day of dosing (Day 1)
* Requiring concomitant therapy with prohibited medications
* Body mass index (BMI) <18 kg/m2 or ≥ 40 kg/m2
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including subjects with <3 excised basal cell carcinomas)
* History of a diagnosis of drug or alcohol dependency or abuse within approximately the last 3 years
* Any condition possibly affecting drug absorption (e.g., gastrectomy, gastroplasty, fundoplication, any type of bariatric surgery, vagotomy, or bowel resection)
* Recent history of stroke or transient ischemic attack (within 6 months prior to Screening) not due to trauma, repaired vascular malformation, or aneurysm
* Screening systolic blood pressure (SBP) >160 mm Hg or a diastolic blood pressure (DBP) >90 mm Hg
* QTc interval >450 milliseconds in males, >470 milliseconds in females
* Breastfeeding
* Treatment with an investigational drug or biologic within 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion
* Blood donation within 56 days or plasma donation within 7 days prior to dosing
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the subject inappropriate for entry into this trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2015-08-07 (Actual); Study Completion 2015-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selwyn Spangenthal, Principal Investigator — American Health Research
Locations (1):
- American Health Research, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefapixant: Gefapixant oral tablets (150 mg) administered as a single dose gefapixant: gefapixant oral tablet (150 mg administered as three 50 mg tablets) - single dose only
Period: Overall Study
Arm/Group | Gefapixant
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gefapixant
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
BP [Mean (Full Range); unit: mmHg] — Blood Pressure
  mmHg
    Mean Baseline Systolic BP | 122 [100 to 132]
    Mean Baseline Diastolic BP | 77 [60 to 92]

OUTCOME MEASURES:

1. Primary Outcome: Effect of Gefapixant on BP
Description: BP data will be summarized using descriptive statistics
Time Frame: 6 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Gefapixant
Number analyzed (Participants) | 6
units on a scale
  Mean Systolic BP at 6 hrs | 122 [90 to 142]
  Mean Diastolic BP at 6 hrs | 76 [56 to 96]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Gefapixant
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant (N=6)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Hypogeusia (Nervous system disorders) | 3 (4)
Pain (General disorders) | 1 (1)
Feeling Hot (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Local Swelling (General disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
60 days prior to the submission of any results, the PI shall submit to SPONSOR any proposed PUBLICATION, which period may be extended for an additional 30 days if requested by SPONSOR. If any Confidential Information should be redacted or patent applications relating to an Invention should be filed prior to PUBLICATION, then PUBLICATION will be delayed until patent application has been filed. Delay of a PUBLICATION shall not exceed 24 months from the date of such notice to the PI.